CLINICAL TRIAL: NCT04580316
Title: Active/Passive Parental Presence Influences Behavior of Preschoolers With Different Intelligence and Fear Levels in the Dental Setting: Randomized Clinical Trial
Brief Title: Parental Presence and Preschoolers' Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dina Youssef Attia, Assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Parent active/passive presence
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Parent-Child Relations; Dental Fear
Keywords: Dental fear; Intelligence quotient; Preschool children; Parental technique; Behavior modification

STUDY DESIGN:
Masking Description: Only biostatistician was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 75 children were managed during intervention using Parental Active Presence.
  Interventions: Behavioral: Parental active presence
- control group (Placebo Comparator): 75 children were managed with passive parent presence.
  Interventions: Behavioral: Parent passive presence

INTERVENTIONS:
Behavioral: Parental active presence — The parents were allowed to stand close to their children, do handholding, eye contacting and help in explaining the dentist's instructions.
  Arms: Experimental group
Behavioral: Parent passive presence — Parents were instructed to sit silently in the dental clinic behind the patient with no eye contact, and without a spoken word only to reassure their children
  Arms: control group

SUMMARY:
Purpose: This study aimed to assess the effect of parental active/passive presence technique (PAP/PPP) on the overall behavior of preschool children with different intelligence and fear levels.

Methods: This randomized controlled trial recruited 150 healthy children, 3-6 years old, with no history of previous dental pain/treatment, IQ level ≤70 to ≤110. After sample collection, in the first visit, children were stratified according to their Intelligence Quotient into 3 equal groups (high, average, low) in which each group was further equally and randomly divided into 2 sub-groups (test and control). In the second visit, before intervention with preventive measures, dental fear was assessed using facial image scale. During intervention, the control sub-groups were managed using PPP technique, while the test sub-groups were managed using PAP technique. Overall behavior was assessed using Frankl behavior rating scale at the end of the 2nd visit. Data was analyzed using chi-square test and logistic regression analysis.

Results: The PAP technique had significantly higher odds of positive behavior than the PPP technique (P=0.002).

Conclusions: Children with low intelligence showed higher dental fear and negative behavior in the dental setting. PAP technique had significant positive effect on the children's overall behavior with different fear and intelligence levels.

DETAILED DESCRIPTION:
The design of the study was a randomized controlled clinical trial with an allocation ratio of 1:1. Children enrolled in this study were stratified based on their IQ into three groups; high, average and low IQ groups. In each of these three groups, children were randomly and equally allocated into study and control subgroups. Thus, this study included 6 subgroups.

- Visual Screening and History taking were carried out to identify children who fulfilled the inclusion criteria. Parental meeting was also conducted to explain the child entire research plan.

The children were recruited from the Outpatient clinic of Pediatric Dentistry Department in Faculty of Dentistry at Alexandria University.

The IQ test for each selected child took place in a quiet closed room (special need clinic). The preventive measures were applied in the pediatric clinic of the department.

- Interventions

In the first visit, children who fulfilled the inclusion/ exclusion criteria were evaluated by IQ test then divided into 3 equal groups (50 children) according to their level of intelligence IQ as follows:

1. High IQ Children group (HIQ): with score of (110 and above)
2. Average IQ Children (AIQ): with score of (90-109)
3. Low IQ Children (LIQ)(with the normal intelligence range): with score of (70-89) In the second visit, fear was measured in each group followed by random allocation into test and control subgroups and then the implementation of the intervention.

   * In each group (50 children), 25 children in subgroup S (study group) were managed using Parental Active Presence (PAP) technique, while the other 25 children in subgroup C (control group) were managed using Parental Passive Presence (PPP) technique. Parental Active / Passive Presence technique was accompanied with Tell-Show-Do (TSD) Technique (Addelston, 1959). During this management, dental preventive measures were applied.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 3-6 years (the preoperational stage) (Piaget, 1954; 1966).
2. Patients with no history of previous dental treatment and no history of dental pain.
3. Patients with at least one sound quadrant for sealant application.
4. Patients IQ level should be in the normal intelligence range.

Exclusion Criteria:

1. Multiple dental problems with pain.
2. History of previous dental therapy
3. History of medical and psychological problems
4. Any degree of intellectual disability

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Overall Behavior | 1 month
  Frankl's Behavior Rating Scale (FBRS) (Frankl, Shiere and Fogels, 1962) At the end of the second visit, after the application of preventive measures, each child overall behavior in each group was evaluated according to Frankl's Behavior Rating Scale (FBRS). It is a four group scale used to assess and evaluate the behavior of a child starting from Rating no. 1 (- -) with the most negative child behavior to Rating no. 4 (++) with the most positive child behavior.
Fear Measure | 1 month
  Facial Image Scale (FIS) (Buchanan and Niven, 2002) to account for fear state and is entered into the analysis as a confounder.
  Dental fear was measured in the second visit by administration of Facial Image Scale (FIS). This measurement was done to every child in each group before the start of dental treatment. It is comprised of a row of five faces ranging from very happy face to very unhappy one. Children were asked to point at which face they feel most like at that moment. The face is scored by giving a value of one to the most positive affect face and five to the most negative affect face. The faces with 1 and 2 indicated a low dental fear , while the faces with the value of 4 and 5 indicated high dental fear

CONTACTS AND LOCATIONS:
Overall Officials: Karin M. Dowidar, PhD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We will share the study protocol
Supporting Information: Study Protocol
Time Frame: After 1 month and for 1 year
Access Criteria: Request access

REFERENCES:
- [Background] Shetty RM, Pashine A, Jose NA, Mantha S. Role of Intelligence Quotient (IQ) on anxiety and behavior in children with hearing and speech impairment. Spec Care Dentist. 2018 Jan;38(1):13-18. doi: 10.1111/scd.12264. Epub 2018 Jan 4. PMID 29314150
- [Background] Piira T, Sugiura T, Champion GD, Donnelly N, Cole AS. The role of parental presence in the context of children's medical procedures: a systematic review. Child Care Health Dev. 2005 Mar;31(2):233-43. doi: 10.1111/j.1365-2214.2004.00466.x. PMID 15715702
- [Derived] AlDhelai TA, Khalil AM, Elhamouly Y, Dowidar KML. Influence of active versus passive parental presence on the behavior of preschoolers with different intelligence levels in the dental operatory: a randomized controlled clinical trial. BMC Oral Health. 2021 Aug 28;21(1):420. doi: 10.1186/s12903-021-01781-z. PMID 34454468